CLINICAL TRIAL: NCT00001995
Title: A Double-Blind Randomized Clinical Trial of a Rifabutin Regimen in the Treatment of Mycobacterium-Avium Complex (MAC) Bacteremia in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 048C; CS 087065
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-11

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Rifabutin

INTERVENTIONS:
Drug: Rifabutin

SUMMARY:
To determine if a drug regimen containing rifabutin will eradicate or decrease the numbers of Mycobacterium avium complex (MAC) organisms in blood, improve the symptoms associated with MAC infection, and increase survival in patients with AIDS. To assess the safety of the drug regimen.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Didanosine (ddI).

Patients must have the following:

* Diagnosis of AIDS as defined by the CDC.
* Blood cultures positive for Mycobacterium avium complex or for acid-fast bacilli (AFB).
* Provide written informed consent.

Prior Medication:

Allowed:

* If receiving zidovudine (AZT) or ddI must be taking the medication for at least 4 weeks prior to study entry.
* Required:
* Antipneumocystis prophylactic therapy for at least 4 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Known hypersensitivity to any of the study drugs.

Concurrent Medication:

Excluded:

* Other therapy for mycobacterial disease.

Patients with the following are excluded:

* Known hypersensitivity to any of the study drugs.

Prior Medication:

Excluded within 4 weeks:

* Therapy for mycobacterial disease.
* Antiretroviral drugs, other than zidovudine (AZT) or ddI.
* Investigational drugs, other than ddI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Maricopa County Med Ctr, Phoenix, Arizona
  - Bay Harbor Hosp, Harbor City, California
  - Ctr for Special Immunology, Irvine, California
  - Southwest Community Based AIDS Treatment Group - COMBAT, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - HIV Research Group, San Diego, California
  - Davies Med Ctr, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Mem Hosp Hollywood, Hollywood, Florida
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Infectious Disease Research Consortium of Georgia, Atlanta, Georgia
  - Dr Frank Rhame, Minneapolis, Minnesota
  - Research Med Ctr, Kansas City, Missouri
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Nassau County Med Ctr, East Meadow, New York
  - Chelsea Village Med Ctr / Saint Vincent's Hosp, New York, New York
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Milwaukee County Med Complex, Milwaukee, Wisconsin

REFERENCES:
- [Background] Dautzenberg B, Castellani P, Pellegrin JL, Vittecoq D, Truffot-Pernot C, Pirotta N, Sassella D. Early bactericidal activity of rifabutin versus that of placebo in treatment of disseminated Mycobacterium avium complex bacteremia in AIDS patients. Antimicrob Agents Chemother. 1996 Jul;40(7):1722-5. doi: 10.1128/AAC.40.7.1722. PMID 8807071